CLINICAL TRIAL: NCT03062670
Title: Team-Based Delivery of Care in Outpatient Settings: An Experimental Investigation
Brief Title: Team-Based Delivery of Care in Outpatient Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David R. Rushlow, Assistant Professor of Family Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-010146
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retreat (Experimental): A full day off-site training session
  Interventions: Other: Retreat
- Control (No Intervention): Care teams normal process

INTERVENTIONS:
Other: Retreat — Full day off-site training session
  Arms: Retreat

SUMMARY:
Through this research we intend to evaluate whether a team-based care delivery approach using daily huddles is effective in improving caregiver and patient outcomes in primary care setting. This approach is expected to not only lead to effective primary care delivery outcomes, but also result in greater team morale, reduced burnout, and a higher rate of innovation.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old adult
* member of Mayo care team in the Midwest

Exclusion Criteria:

-Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in team cohesion | Change from baseline to 6 months
  Survey with 5 point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: David R Rushlow, MD, Study Director — Mayo Clinic
Locations (10):
- United States (10):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System in Austin, Austin, Minnesota
  - Mayo Clinic Health System in Cannon Falls, Cannon Falls, Minnesota
  - Mayo Clinic Health System in Lake City, Lake City, Minnesota
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Mayo Clinic Health System in Owatonna, Owatonna, Minnesota
  - Mayo Clinic Health System in Red Wing, Red Wing, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System in Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lampman MA, Chandrasekaran A, Branda ME, Tumerman MD, Ward P, Staats B, Johnson T, Giblon R, Shah ND, Rushlow DR. Optimizing Huddle Engagement Through Leadership and Problem Solving Within Primary Care: Results from a Cluster-Randomized Trial. J Gen Intern Med. 2021 Aug;36(8):2292-2299. doi: 10.1007/s11606-020-06487-6. Epub 2021 Jan 26. PMID 33501530
- [Derived] Branda ME, Chandrasekaran A, Tumerman MD, Shah ND, Ward P, Staats BR, Lewis TM, Olson DK, Giblon R, Lampman MA, Rushlow DR. Optimizing huddle engagement through leadership and problem-solving within primary care: A study protocol for a cluster randomized trial. Trials. 2018 Oct 4;19(1):536. doi: 10.1186/s13063-018-2847-5. PMID 30286798